CLINICAL TRIAL: NCT02981758
Title: Accurate Display of Postpartum Hemorrhage Using Triton (ADOPT) - A Retrospective Blinded Cohort Study
Brief Title: Accurate Display of Postpartum Hemorrhage Using Triton (ADOPT)
Acronym: ADOPT
Status: Completed | Type: Observational
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Other Study IDs: Pro2016-0184
Record Dates: First submitted 2016-11-18; First posted 2016-12-05 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Post-partum Hemorrhage (PPH)
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Data Collection Phase 1: All women who had vaginal deliveries between 2010 and 2015 who had a procedure code indicative of transfusion (99.0x) or received a diagnosis suggestive of peripartum hemorrhage (e.g. diagnosis x code 666.xx, 641.x, 645.x, 646.x 674.x).
- Data Collection Phase 2: All women who delivered (vaginally) at HackensackUMC who had blood loss and measured quantitatively by Triton and qualitatively (i.e., EBL) by obstetrician.

SUMMARY:
A comparison of reported estimated blood loss with quantified blood loss in all patients whose medical records indicate Triton was used during their vaginal delivery.

DETAILED DESCRIPTION:
This study is a retrospective blinded cohort trial comprised of two data collection phases. In the first phase data will be collected on all women who had vaginal deliveries between 2010 and 2015 who had a procedure code indicative of transfusion (99.0x) or received a diagnosis suggestive of peripartum hemorrhage (e.g. diagnosis x code 666.xx, 641.x, 645.x, 646.x 674.x). Phase 2 will consist of all women who delivered (vaginally) at HackensackUMC who had blood loss and measured quantitatively by Triton and qualitatively (i.e., EBL) by obstetrician. This will be accomplished by reviewing the records of women who delivered and were discharged within the data collection period.

ELIGIBILITY:
Inclusion Criteria:

* All women who delivered (vaginally) at HackensackUMC who had blood loss and measured quantitatively by Triton and qualitatively (i.e., EBL) by obstetrician.
* All women who had vaginal deliveries between 2010 and 2015 at HackensackUMC who had a procedure code indicative of transfusion (99.0x) or received a diagnosis suggestive of peripartum hemorrhage (e.g. diagnosis x code 666.xx, 641.x, 645.x, 646.x 674.x).

Exclusion Criteria:

* Women who received transfusions unrelated directly to pregnancy (e.g. renal disease, anemia of pregnancy, genetic or viral conditions causing anemia).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All women who delivered (vaginally) at HackensackUMC between 2010 and 2015 who had blood loss during the delivery.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2016-07; Primary Completion 2018-07 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Quantification of blood loss during vaginal deliveries | During labor
  Retrospective Chart Review of blood loss during delivery
Quantification of blood loss during vaginal deliveries | During delivery (intrapartum)
  Retrospective Chart Review of blood loss during delivery
Quantification of blood loss during vaginal deliveries | During immediate postpartum period.
  Retrospective Chart Review of blood loss during delivery

SECONDARY OUTCOMES:
Comparison of quantified blood loss (hemoglobin loss) using the The Triton™ System of mobile imaging with computer vision and learning algorithms compared to estimations of blood loss given by the provider. | During labor
  Retrospective Chart Review of blood loss during delivery
Comparison of quantified blood loss (hemoglobin loss) using the The Triton™ | During delivery (intrapartum)
  Retrospective Chart Review of blood loss during delivery
Comparison of quantified blood loss (hemoglobin loss) using the The Triton™ | During immediate postpartum period.
  Retrospective Chart Review of blood loss during delivery

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Rubenstein, M.D., Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack University Medical Center, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Al Kadri HM, Al Anazi BK, Tamim HM. Visual estimation versus gravimetric measurement of postpartum blood loss: a prospective cohort study. Arch Gynecol Obstet. 2011 Jun;283(6):1207-13. doi: 10.1007/s00404-010-1522-1. Epub 2010 May 28. PMID 20508942
- [Result] Berg CJ, Harper MA, Atkinson SM, Bell EA, Brown HL, Hage ML, Mitra AG, Moise KJ Jr, Callaghan WM. Preventability of pregnancy-related deaths: results of a state-wide review. Obstet Gynecol. 2005 Dec;106(6):1228-34. doi: 10.1097/01.AOG.0000187894.71913.e8. PMID 16319245
- [Result] Brant HA. Precise estimation of postpartum haemorrhage: difficulties and importance. Br Med J. 1967 Feb 18;1(5537):398-400. doi: 10.1136/bmj.1.5537.398. No abstract available. PMID 5297397
- [Result] Calvert C, Thomas SL, Ronsmans C, Wagner KS, Adler AJ, Filippi V. Identifying regional variation in the prevalence of postpartum haemorrhage: a systematic review and meta-analysis. PLoS One. 2012;7(7):e41114. doi: 10.1371/journal.pone.0041114. Epub 2012 Jul 23. PMID 22844432
- [Result] Centers for Disease Control and Prevention Mortality Data Run (November 17, 2015)
- [Result] D'Alton ME, Main EK, Menard MK, Levy BS. The National Partnership for Maternal Safety. Obstet Gynecol. 2014 May;123(5):973-977. doi: 10.1097/AOG.0000000000000219. PMID 24785848
- [Result] Della Torre M, Kilpatrick SJ, Hibbard JU, Simonson L, Scott S, Koch A, Schy D, Geller SE. Assessing preventability for obstetric hemorrhage. Am J Perinatol. 2011 Dec;28(10):753-60. doi: 10.1055/s-0031-1280856. Epub 2011 Jun 22. PMID 21698554
- [Result] Dildy GA 3rd, Paine AR, George NC, Velasco C. Estimating blood loss: can teaching significantly improve visual estimation? Obstet Gynecol. 2004 Sep;104(3):601-6. doi: 10.1097/01.AOG.0000137873.07820.34. PMID 15339775
- [Result] Duthie SJ, Ven D, Yung GL, Guang DZ, Chan SY, Ma HK. Discrepancy between laboratory determination and visual estimation of blood loss during normal delivery. Eur J Obstet Gynecol Reprod Biol. 1991 Jan 30;38(2):119-24. doi: 10.1016/0028-2243(91)90188-q. PMID 1995380
- [Result] Knight M, Callaghan WM, Berg C, Alexander S, Bouvier-Colle MH, Ford JB, Joseph KS, Lewis G, Liston RM, Roberts CL, Oats J, Walker J. Trends in postpartum hemorrhage in high resource countries: a review and recommendations from the International Postpartum Hemorrhage Collaborative Group. BMC Pregnancy Childbirth. 2009 Nov 27;9:55. doi: 10.1186/1471-2393-9-55. PMID 19943928
- [Result] Patel A, Goudar SS, Geller SE, Kodkany BS, Edlavitch SA, Wagh K, Patted SS, Naik VA, Moss N, Derman RJ. Drape estimation vs. visual assessment for estimating postpartum hemorrhage. Int J Gynaecol Obstet. 2006 Jun;93(3):220-4. doi: 10.1016/j.ijgo.2006.02.014. Epub 2006 Apr 12. PMID 16626718
- [Result] PRITCHARD JA. CHANGES IN THE BLOOD VOLUME DURING PREGNANCY AND DELIVERY. Anesthesiology. 1965 Jul-Aug;26:393-9. doi: 10.1097/00000542-196507000-00004. No abstract available. PMID 14313451
- [Result] Rath WH. Postpartum hemorrhage--update on problems of definitions and diagnosis. Acta Obstet Gynecol Scand. 2011 May;90(5):421-8. doi: 10.1111/j.1600-0412.2011.01107.x. PMID 21332452
- [Result] Royal College of Obstetrician and Gynaecologists. (2011). Postpartum hemorrhage: prevention and management. Retrieved May2, 2016 from http://www.cedepap.tv/GPC17.pdf
- [Result] Schorn MN. Measurement of blood loss: review of the literature. J Midwifery Womens Health. 2010 Jan-Feb;55(1):20-7. doi: 10.1016/j.jmwh.2009.02.014. PMID 20129226
- [Result] Stafford I, Dildy GA, Clark SL, Belfort MA. Visually estimated and calculated blood loss in vaginal and cesarean delivery. Am J Obstet Gynecol. 2008 Nov;199(5):519.e1-7. doi: 10.1016/j.ajog.2008.04.049. Epub 2008 Jul 17. PMID 18639209
- [Result] Joint Commission on Accreditation of Healthcare Organizations, USA. Preventing maternal death. Sentinel Event Alert. 2010 Jan 26;(44):1-4. No abstract available. PMID 20183946
- [Result] Toledo P, McCarthy RJ, Hewlett BJ, Fitzgerald PC, Wong CA. The accuracy of blood loss estimation after simulated vaginal delivery. Anesth Analg. 2007 Dec;105(6):1736-40, table of contents. doi: 10.1213/01.ane.0000286233.48111.d8. PMID 18042876
- [Result] WHO. Trends in maternal mortality 1990 -2008 estimates developed by WHO, UNICEF, UNFPA and The World Bank, World Health Organization 2010 Annex 1 http://whsqibdoc.who.int/publications2010/9789241500265
- [Result] Zelop CM. Postpartum hemorrhage: becoming more evidence-based. Obstet Gynecol. 2011 Jan;117(1):3-5. doi: 10.1097/AOG.0b013e318202ec9a. No abstract available. PMID 21173639